CLINICAL TRIAL: NCT05471089
Title: Non-invasive Radiofrequency Diathermy and Supervised Therapeutic Exercise in Patellofemoral Pain Syndrome. A Single Blind Randomized Controlled Trial With a Six-month Follow-up
Brief Title: Long-term Effects of the Addition of Diathermy by Emission of Radiofrequency to Therapeutic Exercise in Patellofemoral Pain Syndrome Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jaén (Other)
Responsible Party: Principal Investigator, Alfonso Javier Ibáñez-Vera, Professor of the Department of Health Sciences, University of Jaén
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PFPS 3
Record Dates: First submitted 2022-07-11; First posted 2022-07-22 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Patellofemoral Pain Syndrome; Patellofemoral Pain; Patello Femoral Syndrome
Keywords: knee pain; electrophysical agents
MeSH Terms: conditions — Patellofemoral Pain Syndrome | interventions — Exercise Therapy

STUDY DESIGN:
Intervention Model Description: Double-blind Randomized Controlled Trial
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants were unaware of the treatment group. Researchers in charge of assessment were blinded. Investigator in charge of data analysis was blinded about treatments. Only care providers known about the different treatments
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Application of radiofrequency diathermy in addition to the exercises protocol same Exercise protocol than control group. Ten sessions of treatment were applied: daily the first week (Monday to Friday), three the second week (Monday, Wednesday, Friday) and two the last week (Monday and Thursday)
  Interventions: Device: Diathermy by emission of Radiofrequency; Other: Therapeutic exercise
- Control (Active Comparator): Exercise protocol consisting of: eccentric and concentric strengthening of quadriceps (three squat series of 20 repetitions), hamstrings (three series of 20 seconds performing the bridge exercise), gluteus medius (three series of 20 seconds performing the clam exercise), gastrocnemius and soleus (three series of stretching exercises for 1 minute each). These exercises will be performed along 20 minutes approximately with a minute of rest between each exercise series, never exceeding 3mm in VAS. Participants have to assist to a local facility center to be supervised at doing the exercises daily (from Monday two Friday) along three weeks.
  Interventions: Other: Therapeutic exercise

INTERVENTIONS:
Device: Diathermy by emission of Radiofrequency — Applied only to experimental group
  Arms: Experimental
Other: Therapeutic exercise — Applied to both arms/groups

SUMMARY:
Introduction: the management of Patellofemoral Pain (PFP) is focused on therapeutic exercise (TE) to improve muscle strength and motor control. Recent studies suggest that the addition of radiofrequency diathermy (RFD) obtain greater short-term improvements in knee pain than TE alone. As there is no follow up data, the aim of this research is to assess the long-term effects of adding RFD to TE on pain, function and quality of life on PFP patients.

Methods: a single-blind randomized controlled trial will be conducted. Participants diagnosed of PFP will be allocated in either a TE group or a RFD+TE one. Sociodemographic data, knee pain, and lower limb function will be collected. Each group will performed 20 min of daily knee and hip supervised TE along three weeks with the addition of ten sessions of RFD for the RFD+TE group.

ELIGIBILITY:
Inclusion Criteria:

* Subjects between 30 and 50 years old without radiological findings of osteoarthritis.
* Subjects referring during the last month almost three points of pain in the anterior surface of knee measured with Visual Analogue Scale.

Exclusion Criteria:

* Subjects with contraindications for the treatment with radiofrequency diathermy (tumors, use of pacemakers or any other implanted electronic device, thrombophlebitis or deep venous thrombosis, pregnancy, fever, active tuberculosis, infections and rheumatoid arthritis).
* Subjects who have received corticoid or hyaluronic acid or platelet-rich plasma injections treatment in the knee.

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 86 (Actual)
Dates: Start 2022-07-26 (Actual); Primary Completion 2023-02-10 (Actual); Study Completion 2023-02-10 (Actual)

PRIMARY OUTCOMES:
Knee pain | Baseline
  Pain measured with Visual Analogue Scale
Knee pain | At three weeks
  Pain measured with Visual Analogue Scale
Knee pain | Through study completion, an average of 6 months
  Pain measured with Visual Analogue Scale
Knee function | Baseline
  Knee function measured with "Lower Extremity Functional Scale"
Knee function | At three weeks
  Knee function measured with "Lower Extremity Functional Scale"
Knee function | Through study completion, an average of 6 months
  Knee function measured with "Lower Extremity Functional Scale"
Knee function | Baseline
  Knee function measured with "Kujala score"
Knee function | At three weeks
  Knee function measured with "Kujala score"
Knee function | Through study completion, an average of 6 months
  Knee function measured with "Kujala score"

CONTACTS AND LOCATIONS:
Locations (1):
- Centro de Salud San José de la Rinconada, Seville, Spain

IPD SHARING:
Plan to Share IPD: No